CLINICAL TRIAL: NCT06349395
Title: The Effect of Mindfulness-Based Stress Reduction Training Before Mastectomy on Postoperative Pain in Early Period
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Rabia Buse Ayyildiz, Principal Investigator, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NisantasiU
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-03

CONDITIONS: Pain Management
Keywords: MBSR; surgical nursing; pain management; fear of movement; mastectomy
MeSH Terms: conditions — Agnosia; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: 2 parallel groups randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): The study conducted an online eight-session mindfulness-based stress reduction (MBSR) program for its intervention group, with each session lasting about two hours. Daily exercise adherence was monitored via phone. The control group received no intervention but followed standard hospital protocols, with an offer for MBSR training post-study.
  Interventions: Other: MBSR surgical nursing care
- controls(control group) (No Intervention): No intervention was provided to the control group; these participants were evaluated following the routine hospital treatment protocol. Participants who wished to receive MBSR training were offered the opportunity to do so after the completion of the study.

INTERVENTIONS:
Other: MBSR surgical nursing care — This study delivered an eight-session mindfulness-based stress reduction (MBSR) program online to its intervention group, each lasting about two hours, incorporating daily exercises monitored via phone. The evaluation of MBSR's effectiveness focused on postoperative pain at 6, 12, 18, and 24 hours after surgery and assessed fear of movement before starting arm exercises on the 5th day post-mastectomy. This approach provided a detailed examination of MBSR's role in pain and movement fear management, highlighting its potential as a preoperative care component for breast cancer patients.
  Arms: interventional

SUMMARY:
This research aims to investigate the effect of mindfulness-based stress reduction training given before mastectomy on postoperative early period pain and the fear of movement caused by pain. According to the World Health Organization, 18.1 million new cancer diagnoses are made each year, with breast cancer being the most common type among women, accounting for 24.2% of all cancers diagnosed. In Turkey, the incidence of breast cancer was determined as 22,345 in 2018. Breast cancer significantly affects women's quality and length of life. Surgical intervention is the most commonly chosen treatment method for cases of localized breast cancer. Pain and limited movement are among the most common problems encountered after surgery. Non-pharmacological methods have been shown to be effective in pain management, with the mindfulness-based stress reduction technique being one of these methods. This technique is described as an effective treatment for conditions such as pain, depression, and addiction, with high levels of mindfulness being associated with greater self-esteem, optimism, and empathy, whereas low levels of mindfulness are linked to depression, anxiety, chronic pain, and acute pain.

DETAILED DESCRIPTION:
This research aims to explore the effectiveness of mindfulness-based stress reduction (MBSR) training, delivered through an eight-session program prior to mastectomy, in alleviating postoperative pain-a critical challenge in breast cancer treatment. Recognizing the substantial impact of breast cancer on women's quality of life and the limitations of traditional pharmacological approaches to pain management, this study proposes a non-pharmacological intervention. By employing an experimental design, it investigates whether preoperative MBSR training can lead to a significant reduction in pain levels among patients undergoing mastectomy, compared to those who do not receive such training. The hypothesis suggests that mindfulness training, by fostering higher levels of mindfulness, may improve pain management, thereby enhancing patient outcomes and suggesting a potential shift towards incorporating holistic preparatory training in standard preoperative protocols. This approach aims to contribute to the evolving landscape of pain management strategies in breast cancer care, emphasizing patient-centered and integrative treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Verbally and in writing agreed to participate in the study after being informed about the research, Are aged 18 and over, Can read, write, and speak Turkish, understand the provided information, and have no issues with verbal communication, Do not have any physical issues that would prevent participation in mindfulness-based stress reduction training, Have not previously received mindfulness-based stress reduction training, Underwent surgery with general anesthesia, Had arterial blood pressure, pulse, oxygen saturation, and body temperature within normal limits during and after surgery, Received non-narcotic and consistent analgesic substances postoperatively for pain control, Were administered antibiotics postoperatively with the same active ingredient.

Exclusion Criteria:

* Patients without internet access, Those unable to use the application through which the training is provided or without someone to assist them, Individuals who cannot allocate regular time for the training, Patients with chronic pain during the preoperative period who are using analgesics for treatment, Patients with restricted movement activity before the surgery will not be included

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — being female
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-29 (Estimated); Study Completion 2024-07-29 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | after operation 6.hours, 12 hours, 18 hours, 24 hours
  Pain assessment: Pain scores of patients will be recorded using 0-100 mm Visual Analog Scale (VAS) to grade pain. For VAS; A measured horizontal line will be created, and definitions such as 'no symptoms' and 'severe symptoms' will be written at both ends. The participant will be instructed to mark a point on the line appropriate to the severity of the symptom. Wrist pain values in the resting position will be recorded before and after the 6-week program.
The Tampa Scale of Kinesiophobia | after operation before starting arm exercises (5th day)
  fear of movement (TSK) is a measure used to assess fear of movement/(re)injury. It is often utilized in clinical settings to evaluate the degree to which fear of physical movement and activity due to beliefs of vulnerability to injury affects individuals, particularly those recovering from injury or dealing with chronic pain conditions.The Tampa Scale of Kinesiophobia (TSK) typically has a minimum score of 17 and a maximum score of 68. The scale consists of 17 items, each rated on a 4-point Likert scale ranging from "strongly disagree" (1 point) to "strongly agree" (4 points). Higher scores indicate greater fear of movement or re-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Öztekin, Prof., Study Director — Dogus Universitesi
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No